CLINICAL TRIAL: NCT07231562
Title: The Effect of Mobilization Training Given to Patients Undergoing Lumbar Stabilization Surgery on Postoperative Pain, Anxiety, Kinesiophobia, Fear of Falling, and Mobility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Oğuz Özdemir, Principal Investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SDU-Hemsire-OÖ-001
Record Dates: First submitted 2025-10-01; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Disease; Lumbar Surgery
Keywords: Lumbar region; kinesiophobia; mobilization; nursing care and education; perioperative period
MeSH Terms: conditions — Disease; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: an intervention group that would receive mobilization training and a control group that would not receive training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): A group of 30 patients who will receive training on mobilization by watching videos and brochures using virtual reality glasses during the preoperative period (Intervention group).
  Interventions: Other: The group that will receive mobilization training using virtual reality glasses and brochures
- control group (No Intervention): A group of 30 patients who did not receive any video or brochure training other than the routine mobilization process during the preoperative period, and whose differences were examined and compared with those in the intervention group (control group).N

INTERVENTIONS:
Other: The group that will receive mobilization training using virtual reality glasses and brochures — A group of 30 patients who will receive training on mobilization by watching videos and brochures using virtual reality glasses during the preoperative period (Intervention group).
  Other Names: the group to be given mobilization training
  Arms: intervention group

SUMMARY:
In this study, the researcher will examine the effects of preoperative mobilization training (video viewing with VR glasses and brochure methods) given to patients undergoing surgery in the lumbar region on pain, anxiety, fear of movement, fear of falling, and mobility levels in the postoperative period, using specific scales.

DETAILED DESCRIPTION:
Conditions requiring surgical intervention in the lumbar region include various pathological conditions such as lumbar disc herniation, spinal cord tumors, traumatic spinal injuries, and spinal stenosis. Surgical interventions such as stabilization, fusion, laminectomy, and discectomy are commonly performed for these conditions. The study is a randomized controlled comparative study. The study sample will consist of patients admitted to the Neurosurgery-I and Neurosurgery-II clinics of Eskişehir City Hospital before surgery and transferred back to the clinic after surgery. The study sample is planned to include 60 patients in the intervention group and 60 in the control group. Pre-test data will be collected in the preoperative period from patients in the intervention and control groups who agreed to participate in the study in accordance with the informed consent form and gave their consent using the Informed Consent Form, the Patient Information Form, the State-Trait Anxiety Scale, the Tampa Kinesiophobia Scale, the Likert-Type Fear of Falling Scale, the Visual Analog Scale, the Patient Mobility Scale, and the Observer Mobility Scale. Afterwards, patients in the intervention group will be trained on mobilization by watching a video using VR headsets and using a brochure. Patients in the control group will not receive any video or brochure training other than during the routine mobilization process in the ward. The brochure given to the intervention group will include mobilization and information included in the video viewing using VR headsets and will be given to patients so they can open and read it at any time. During the first mobilization of patients in the intervention and control groups, a "Patient Information Form" will be filled out before mobilization. Data will be collected again using the "State-Trait Anxiety Scale," "Tampa Kinesiophobia Scale," "Likert-Type Fear of Falling Scale," and "Visual Analog Scale." Patients in the intervention group will then be mobilized appropriately using a video and brochure training program shown through virtual reality glasses regarding the mobilization steps. Patients in the control group will be mobilized using the mobilization steps routinely performed in the ward. After the initial mobilization of patients in both groups, data will be collected and recorded again using the "Visual Analog Scale," "Patient Mobility Scale," and "Observer Mobility Scale." As a posttest, before the final mobilization of patients in the intervention and control groups before discharge, they will complete the "Patient Information Form," "State-Trait Anxiety Scale," and "Tampa Kinesiophobia Scale." Post-test data will be collected using the "Likert-Type Fear of Falling Scale," "Visual Analog Scale," and "Visual Analog Scale." Post-test data will be collected and recorded 5-10 minutes after mobilization is achieved using the "Visual Analog Scale," "Patient Mobility Scale," and "Observer Mobility Scale." Data will be collected face-to-face by the researchers. Ethics committee approval, Turkish Medicines and Medical Devices Agency (TİTCK), and institutional permissions have been obtained for the study. Patients will also provide informed consent in accordance with the Informed Consent Form. Statistical analyses will be performed using computer software using numbers, percentages, means, standard deviations, t-tests, and chi-square tests.

ELIGIBILITY:
İnclusion Criteria

* The patient must be over 18 years of age
* Participate in the study voluntarily,
* Be undergoing lumbar surgery for the first time
* Be undergoing lumbar stabilization surgery
* Be oriented to person, place, and time
* Not have taken any oral or parenteral analgesic medication other than the routine treatment ordered before mobilization
* Have no restrictions (physical disability, etc.) that would prevent mobilization,
* Be able to understand and speak Turkish
* Have no vision or hearing problems,
* Have no psychiatric illness, ağrı var
* Be in ASA 1 or 2,
* Patients planned to be included in the intervention and control groups must not be in the same rooms.

Exclusion Criteria

* Having a neurological (such as dementia/Alzheimer's) or psychiatric (such as schizophrenia) medical diagnosis that affects cognitive status.
* Having a chronic pain disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale (TKS) | eight months
  The TSK is a 17-question scale developed to determine the level of injury/re-injury and fear-avoidance processes associated with activities. The scale is scored using a four-point Likert scale: "1 = Strongly Disagree," "2 = Disagree," "3 = Agree," and "4 = Strongly Agree." The minimum score on the scale is 17, while the maximum score is 68.
Patient Mobility Scale-HHO | eight months
  The Patient Mobility Scale consists of eight items and four subscales: turning from side to side in bed, sitting at the edge of the bed, standing at the edge of the bed, and walking in the patient's room. The level of pain and difficulty experienced is assessed using a 15-cm visual analog with verbal statements listed below the scale. The numerical value of the degree of pain and difficulty is determined by measuring the distance between the patient's mark on the scale and "0" using a calibrated ruler (no pain, some pain, moderate pain, a lot of pain, the worst pain I can imagine/very easy, easy, a little difficult, difficult, very difficult). The lowest and highest scores for each item range from 0 to 15, and the total scale score ranges from 0 to 120.

SECONDARY OUTCOMES:
Observer Mobility Scale-GHÖ | eight months
  The Observer Mobility Scale provides global observations of four subscales: turning from side to side in bed, sitting at the edge of the bed, standing up at the edge of the bed, and walking in the patient's room. Each subscale is scored from 1 to 5, with a score of 1 indicating that the patient independently performs the movement without verbal prompting or physical assistance, and a score of 5 indicating that the patient is unable to perform the movement despite verbal prompting or physical assistance. The lowest possible score on the scale is 4, and the highest is 20.
Visual Anolog Skala-VAS | eight months
  This scale is a 10-cm ruler, with a minimum value of 0 on one end and a maximum value of 10 on the other. The patient is explained that there are two extremes, and that they are free to mark any point between them that matches the intensity of their pain. The distance between the onset of "no pain" and the point marked by the patient is measured in centimeters and recorded.
State and Trait Anxiety Scale | eight months
  State Anxiety Scale (items 1-20):
  * Determines an individual's current anxiety level.
  * Contains 10 direct and 10 reversed statements.
  * Direct and reversed statements are scored differently.
  * Calculation: (Total direct statements - Total reverse statements) + 50.
  Trait Anxiety Scale (items 21-40):
  * Measures an individual's general tendency to anxiety.
  * Contains 13 direct and 7 reversed statements.
  * Calculation: (Total direct statements - Total reverse statements) + 35.
  * Score Range: Both scales yield scores between 20-80.
  * 0-19: No anxiety
  * 20-39: Mild anxiety
  40-59: Moderate anxiety
  60-79: Severe anxiety (60 and above requires professional help).
Likert-Type Fear of Falling Scale | eight months
  The Likert-type scale includes the question, "Are you afraid of falling?" and the answers, "I am very afraid, I am moderately afraid, I am slightly afraid, and I am not afraid at all." The scale consists of a minimum of one (1) and a maximum of four (4) points (12). The scale will be used in this study to determine the level of fear of falling in patients.
Patient Information Form | eight months
  It was developed by the researcher based on literature. It includes questions regarding the patients' age, gender, height, weight, marital status, and educational background. It also includes questions regarding clinical characteristics such as the presence of chronic disease, history of preoperative activity limitation, and history of previous spinal surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz ÖZDEMİR, Principal Investigator — Suleyman Demirel University
Locations (1):
- Eskişehir Şehir Hastanesi, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not want to share the IPD without any justification.

REFERENCES:
- See also: Ko, SY, Leung, DY, & Wong, EM (2019). Effects of easy-listening music intervention on satisfaction, anxiety, and pain in patients undergoing colonoscopy: a pilot randomized controlled trial. Clinical interventions in aging, 14 , 977-986. — https://doi.org/10.2147/CIA.S207191
- See also: Öztaş B, Kara B, Zengin H, Güçlü A, On B. The Effect of Simulation Laboratory Education on Intravenous Catheterization Skills of Nursing Students. HUHEMFAD. 2022;9(1):17-23. — https://doi.org/10.31125/hunhemsire.1101859
- See also: Vlaeyen JW, Kole-Snijders AM, Boeren RG, Van Eek H. Fear of movement/(re)injury in chronic low back pain and its relation to behavioral performance. Pain. 1995; 62(3): 363-372. — https://pubmed.ncbi.nlm.nih.gov/8657437/
- See also: Biçer B. The effect of fear of falling on mobilization-induced fear of movement and fall risk in patients undergoing surgery. Dokuz Eylül University, Institute of Health Sciences, Unpublished Master's Thesis, İzmir, (Assoc. Prof. Dr. Özlem Bilik), 2019; — https://tez.yok.gov.tr/UlusalTezMerkezi/tezDetay.jsp?id=-tBkg4xjGrh-tKJmmKpL5w&no=tMPVR0b4WsdporjxFt3nWg
- See also: Çilingir D, Uzun Şahin C. I woke up early and went ahead: Evidence-based practices in postoperative planned mobilization. Gürsoy A, editor. Evidence-Based Practices in Perioperative Nursing. 1st ed. Ankara: Türkiye Clinics; 2020. p.35-9 — https://www.turkiyeklinikleri.com/article/tr-erken-kalktim-yol-aldim-postoperatif-planli-mobilizasyonda-kanita-dayali-uygulamalar-89613.html
- See also: Geçit S, Özbayır T. Protocol and nursing for accelerating recovery after spinal cord surgery. Özbayır T, editor. Protocol and nursing for accelerating recovery after surgery. 1st ed. Ankara: Türkiye Clinics; 2021. p.83-9. — https://www.turkiyeklinikleri.com/article/tr-spinal-kord-cerrahisi-sonrasi-yilesmenin-hizlandirilmasi-protokolu-ve-hemsirelik-94301.html
- See also: Mahmudova R, Dönmez YC. Investigation of factors affecting the ability of patients to stand up after surgery. Turkish Clinics Journal of Nursing Sciences 2019; 11(1). — https://www.turkiyeklinikleri.com/article/tr-ameliyat-sonrasi-hastalarin-ayaga-kalkma-durumlarini-etkileyen-faktorlerin-ncelenmesi-83625.html